CLINICAL TRIAL: NCT00211692
Title: Prospective Randomized Pilot Study of Daily Consensus Interferon (CIFN) and Ribavirin for 52 Wks vs Extended Duration 72 Wks Based on Virologic Response for the Initial Treatment of Difficult-to-treat Patients With Chronic HCV Genotype 1
Brief Title: Hepatitis C Treatment Naive Genotype 1 Consensus Interferon Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Center for Veterans Research and Education (Other); InterMune (Industry); Kadmon Corporation, LLC (Industry); US Department of Veterans Affairs (U.S. Federal Agency); San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Samuel B. Ho, Staff Physician, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MVRI001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; interferon alfa; ribavirin; interferon alfacon-1; antiviral therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — interferon alfacon-1; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A consensus interferon+rbv 52 wks (Active Comparator): Daily CIFN (15 mcg/day SQ) and RBV (1-1.2 g/d PO) given 52 weeks (group A)
  Interventions: Drug: consensus interferon (Interferon Alfacon-1) and ribavirin; Drug: Consensus Interferon alfa (CIFN) and ribavirin
- Group B CIFN variable duration (Experimental): CIFN (15 mcg/day SQ) and RBV (1-1.2 g/d PO) given for 52-72 weeks (from time of viral response +48 weeks) (group B)
  Interventions: Drug: Consensus Interferon alfa (CIFN) and ribavirin

INTERVENTIONS:
Drug: consensus interferon (Interferon Alfacon-1) and ribavirin — CIFN (15 mcg/day SQ) and RBV (1-1.2 g/d PO) given for either 52 weeks (group A, n = 33) or 52-72 weeks (from time of viral response +48 weeks) (group B)
  Other Names: interferon alfacon-1
  Arms: Group A consensus interferon+rbv 52 wks
Drug: Consensus Interferon alfa (CIFN) and ribavirin — CIFN (15 mcg/day SQ) and RBV (1-1.2 g/d PO) given for either 52 weeks (group A, n = 33) or 52-72 weeks (from time of viral response +48 weeks) (group B)
  Other Names: interferon alfacon-1

SUMMARY:
Data have suggested that consensus interferon (CIFN) has greater antiviral activity in vitro compared with interferon alfa-2a or alfa-2b. Several clinical studies also suggest that CIFN has greater antiviral activity in patients with genotype 1 hepatitis C infection, particularly if given as a daily injection. These data indicate that the use of a regimen of daily CIFN and ribavirin will lead to greater virologic response rates compared with pegylated interferon alfa-2b and ribavirin in patients with genotype 1 infection, with comparable adverse events. Emerging data indicate that HCV genotype 1 patients with a delayed virologic response to initial therapy may benefit from an extended duration of therapy. Therefore, the goals of this pilot study are to determine the tolerability and efficacy of daily CIFN plus ribavirin when given for 52 weeks or an extended duration of therapy. The target population will consist of "difficult-to-treat" patients, defined as having the following characteristics: genotype 1, a North American patient population, predominantly male gender, and no specific exclusions for pre-existing psychiatric or substance abuse co-morbidities.

DETAILED DESCRIPTION:
Current treatment for hepatitis C is a pegylated interferon alfa plus ribavirin. This treatment is inadequate for patients with HCV genotype 1, since the majority of patients do not respond (termed non-responders) or respond but relapse (termed relapsers) following termination of these treatments. Data from the Veterans Health Administration (VHA) Hepatitis C Registry and community hospitals indicate that the large majority of patients identified with hepatitis C have characteristics associated with a poor treatment response and remain untreated at this time. Data have suggested that consensus interferon (CIFN, CIFN or interferon alfacon-1) has greater antiviral activity in vitro compared with interferon alfa-2a or alfa-2b. Preliminary data indicate that more patients with genotype 1 can respond to CIFN and ribavirin than current standard treatments, due to the fact that approximately 25% of patients who are nonresponders to pegylated interferon and ribavirin may have a sustained response to a regimen of daily CIFN and ribavirin. Furthermore, difficult to treat patients may benefit from a longer duration of therapy than the standard 48 week regimen based on when an initial virologic response to therapy occurs.

Aims: To determine the safety and efficacy of (A) daily CIFN (15 mcg/d sq) and ribavirin (1-1.2 gm/d PO) given for 52 weeks, vs (B) daily CIFN (15 mcg/d sq) and ribavirin (1-1.2 gm/d PO) given for 52 to 72 weeks for treatment-naïve patients with hepatitis C genotype 1, with treatment duration based on the virologic response during the initial 24 weeks.

Methods: Patients who meet eligibility criteria will be stratified by race and randomized to one of two treatment arms, and all patients will have viral kinetics measured by quantitative PCR at weeks 4,8,12,16,20 and 24. Patients in treatment arm A will follow "standard" stopping rules, i.e., if there is not a 2-log drop in viremia by 12 weeks the treatment will be discontinued, otherwise they will all receive 52 weeks of treatment if they also are qualitative PCR negative by week 24. In treatment arm B the patients will be monitored monthly until they have a virologic response (defined as >2 log drop in viral levels from baseline) by quantitative PCR for up to 24 weeks. Once they have a virologic response by quantitative PCR their treatment will be continued for an additional 48 weeks. In both groups, treatment will be stopped if the patients do not become negative for HCV RNA by qualitative PCR by 24 weeks on therapy. A total of 192 patients at up to 10-20 sites will be recruited. The primary endpoint would be the number who achieve a sustained virologic response; secondary endpoints are the percentage of patients who complete therapy, have significant adverse events, and the relationship of early virologic response at each 4 week period between 4 and 24 weeks and those who achieve a sustained virologic response.

Sample size determination: To detect an absolute difference of 20% or more in sustained virologic response between treatment arms A and B; the Log-rank test is performed at the alpha level of .05 and the test is maintained at least 80 percent statistical power; it is estimated that a total of 96 patients in each treatment arm will be required.

Analysis: Univariate and multivariate analysis will be used to determine factors associated with final endpoints. Subgroup analyses will be done based on time to early virologic response and duration of therapy each stratification. The primary and secondary endpoints will be determined on an intention-to-treat basis starting with all patients that receive at least one dose of study medications. The primary and secondary endpoints will also be determined in a per-protocol analysis on those patients who take 80% of the prescribed CIFN and 80% of the prescribed ribavirin for 80% of the time.

Significance: The current initial treatment of pegylated interferon alfa and ribavirin for patients with hepatitis C who are genotype 1 and have other "difficult-to-treat" characteristics is inadequate. The results of this trial are needed to demonstrate the safety and efficacy of two regimens of daily CIFN and ribavirin. Since the large majority of hepatitis C patients in VA and other community hospitals fall into this category, the results of this trial may influence the potential treatments recommended for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic hepatitis C. This is defined as the documentation of the presence of circulating hepatitis C virus by a positive hepatitis C PCR test and a positive HCV genotype test for genotype 1, and a liver biopsy (within the previous 5 years) that is compatible with chronic hepatitis. In the case of patients that have refused liver biopsies a clinical diagnosis of chronic hepatitis C is required.

2. Positive HCV RNA by PCR, Genotype 1, treatment naive 3. Age 18-65 years. 4. Patient must be able to give informed consent. 5. Eligible for interferon alfa and ribavirin-based antiviral treatment:

1. Reconfirmation and documentation that sexually active female patients of childbearing potential are practicing adequate contraception. A urine pregnancy test obtained at entry prior to the initiation of treatment must be negative.
2. Reconfirmation that sexually active male subjects are practicing acceptable methods of contraception during the treatment period and for six months following the last dose of study medication.
3. For patients with cirrhosis or stage 4 fibrosis on liver biopsy, they must have an alpha fetoprotein (AFP) value < 80 ng/mL obtained within 3 months prior to entry. Cirrhotics with an alpha fetoprotein value >30 ng/mL but <80ng/mL may be enrolled after a normal ultrasound or triphasic CT scan within the previous 3 months. Cirrhotics with alpha fetoprotein levels up to 30 ng/ml must have an ultrasound or CT scan within 6 months of enrolling that is negative for hepatocellular cancer. Patients with an AFP > 80 ng/mL may not be enrolled.

5) Compensated liver disease with the following laboratory results at entry:

* Hemoglobin >=to 12 gm/dL for females and >= 13gm/dl for males
* WBC >= 2,000/mm3
* Neutrophil >=1,500/mm3
* Platelets >=75,000/mm3
* Albumin > 3.0 g/dL
* Total bilirubin <2.0
* Serum creatinine < 1.4 mg/dL
* INR <1.8
* If diabetic, must have glycosylated Hgb test that demonstrates adequate control of diabetes in the opinion of the investigator
* TSH within normal limits

Exclusion Criteria:

1. Patient unable or unwilling to participate.
2. Liver disease in addition to chronic hepatitis C (HBsAg positive, autoimmune liver disease, hemochromatosis, PBC, PSC, alpha-1 antitrypsin deficiency, Wilson's disease, etc.)
3. Decompensated liver disease, with history of encephalopathy, variceal bleeding, or ascites or CHILD-PUGH class B or C.
4. Baseline BDI > 19 or current suicidal or homicidal ideation. (Note: if baseline BDI is > 19 pt. will require a psychiatric evaluation and treatment; if deemed stable after this he may be considered according to site PI clinical judgment.)
5. Current substance use disorder (Must be evaluated and demonstrate engagement and compliance with care before they will be eligible).
6. Patients with active or uncontrolled psychiatric disease including patients who have had recent prior severe psychiatric disease (hospitalized) within the last 2 years.
7. Accepted and reasonable exclusion criteria for interferon alfa and ribavirin based treatments:

1) CNS trauma or active seizure disorders requiring medication. 2) Significant cardiovascular dysfunction within the past 12 months 3) Poorly controlled diabetes mellitus (in the opinion of the site PI). 4) Moderate or severe chronic pulmonary disease 5) Clinically significant immunologically mediated disease 6) Hemoglobinopathies (e.g., Thalassemia) or any other cause of hemolytic anemia.

7) Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids.

8) Hypersensitivity to interferon alfa or ribavirin 9) Known anti-HIV positive 10) Clinically significant retinopathy 11) Previous solid organ transplantation 12) Any condition that, in the opinion of the investigator, will prevent the patient from being compliant with study medications or appointments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel B. Ho, M.D., Principal Investigator — US Department of Veterans Affairs

REFERENCES:
- [Result] Ho SB, Aqel B, Dieperink E, Liu S, Tetrick L, Falck-Ytter Y, DeComarmond C, Smith CI, McKee DP, Boyd W, Kulig CC, Bini EJ, Pedrosa MC. U.S. multicenter pilot study of daily consensus interferon (CIFN) plus ribavirin for "difficult-to-treat" HCV genotype 1 patients. Dig Dis Sci. 2011 Mar;56(3):880-8. doi: 10.1007/s10620-010-1504-y. Epub 2011 Jan 11. PMID 21221804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with difficult-to-treat characteristics (78% VA) were enrolled at 7 Veterans Affairs (VA) and 2 community medical centers.
Pre-assignment Details: All eligible patients were randomized and analysis performed using intention to treat.
Groups:
- Group A 52 Weeks Treatment: Daily CIFN (15 mcg/day SQ) and RBV (1-1.2 g/d PO) given 52 weeks (group A)
- Group B Duration Based on Viral Response: CIFN (15 mcg/day SQ) and RBV (1-1.2 g/d PO) given for 52-72 weeks (from time of viral response +48 weeks) (group B)
Period: Overall Study
Arm/Group | Group A 52 Weeks Treatment | Group B Duration Based on Viral Response
Started | 33 | 31
Completed | 33 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A 52 Weeks Treatment | Group B Duration Based on Viral Response | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 31 | 64
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (8.0) | 49.8 (8.8) | 50.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 32 | 28 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 22 | 19 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Would be the Number Who Achieve a Sustained Virologic Response.
Description: Overall sustained virologic response for entire cohort and individual sustained virologic response for different arms of study
Time Frame: 24 weeks after the end of treatment
Population: Convenience sample for pilot trial. Analysis is intention to treat.
Measure: Number; unit: participants
Arm/Group | A (52 Weeks Treatment) | B (Duration Based on Viral Response)
Number analyzed (Participants) | 33 | 31
participants | 11 | 10

2. Secondary Outcome: Number of Participants Discontinuing Early From Study Treatment
Time Frame: through end of study up to 72 weeks
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 64
participants | 26

3. Secondary Outcome: Participants Achieving SVR Categorized by Time of Response
Description: rapid virologic response assessed at 4 weeks, early virologic response assessed at 8-12 weeks, late virologic response assessed at 16-24 weeks
Time Frame: 24 weeks after end of treatment
Population: participants with analyzable data for this outcome
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 42
participants
  rapid virologic response (n=20) | 15
  early virologic response (n=13) | 4
  late virologic response (n=9) | 2

4. Secondary Outcome: Overall Number of Serious Adverse Events
Time Frame: through end of study up to 72 weeks
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 64
participants | 2

ADVERSE EVENTS:
Time Frame: through end of study up to 72 weeks
Description: adverse events were collected for study population as a whole
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 2/64
Other Adverse Events (participants affected / at risk) | 16/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=64)
encephalopathy (Nervous system disorders) | 1 (1)
chest pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=64)
depression/anxiety (Nervous system disorders) | 4 (4)
cellulitis (Skin and subcutaneous tissue disorders) | 3 (3)
other intolerable side effects (General disorders) | 9 (9) — includes fatigue and irritibility

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No